CLINICAL TRIAL: NCT04077502
Title: Repetitive Transcranial Magnetic Stimulation in Treatment of Binge Eating Disorder. A Double Blind Placebo Controlled Study
Brief Title: Repetitive Transcranial Magnetic Stimulation in Treatment of Binge Eating Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Katarína Jaššová, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CharlesUniversityPragueCR
Record Dates: First submitted 2019-08-07; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Binge-Eating Disorder
Keywords: binge eating disorder; craving; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: randomized double blinde and placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants in control group were stimulated by sham repetitive transcranial magnetic stimulation coil. The investigator did not know if the participants were stimulated by real or sham coil. Stimulation was provided by other member of invetigation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stimulated group (Active Comparator): The group stimulated by real coil of rTMS.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- controle group (Sham Comparator): The group stimulated by sham coil of rTMS.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Hypothesis: High-frequency rTMS can significantly reduce craving for food in patients with BED just after the stimulation and also over the one month observation period.

Method: The study was designed as a randomized double blind and placebo controlled one. The active group was stimulated by high-frequency rTMS, with the following stimulation parameters: frequency 10 Hz, 1500 pulses, 107 s inter-train, 100% minimal motor threshold and 10 stimulation session. The control group was stimulated by a sham rTMS coil. The FCQ-S and the FCQ-T questionnaires were used to evaluate the food craving.

DETAILED DESCRIPTION:
The study was realized at Department of Psychiatry First Faculty of Medicine Charles University in Prague and General University Hospital in Prague during 2013 - 2018. The study was approved by the Ethics committee General University Hospital in Prague by a decision dated 23.1.2014, number 1867/13 S-IV (individual research). The study was registered on clinicaltrials.gov.

Two psychiatrists examined each patient who signed up for the study, in order to set the diagnoses. The DSM-5 diagnostic criteria were used for the purpose of the study. The exclusion criteria were mainly based upon contraindications for rTMS such as: a history of epileptic seizure paroxysms, increased intracranial pressure, brain tumor, implanted metal devices in the cranium (except the oral cavity), and any implanted peacemaker or drug pump. Also, patients who were not able to complete 10 sessions of rTMS were excluded for non-compliance. Inclusion criteria were: having BED and being over the age of 18. The study did not account for the hemispherical laterality.

After signing an informed consent form, subjects were included into the study and randomly divided into two groups: one group stimulated by a real rTMS coil (group A - active), and the second (control group), stimulated by a sham rTMS coil (group P - placebo).

Patients were also offered to participate in cognitive behavioral group therapy (CBT) simultaneously with the rTMS treatment. However, the attendance in the CBT was voluntary, and it was not a condition for inclusion into the study.

The study was conceived as randomized double blind placebo controlled clinical study. The randomization was performed by statistics independent of study. The investigators group achieved the study´s double blind characteristics by dividing the roles of the researchers. One author provided the examinations of the patients, CBT, data collection and evaluations of the questionnaires, while a second author administered the stimulations. The control group was "blind" thanks to the use of the sham coil.

Collection of data and statistical analysis Subjects were asked to fill out the set of questionnaires consisting of the EDE-Q (Eating Disorder Examination - Questionnaire), as well as the FCQ-S, and the FCQ-T before the first stimulation session. The EDE-Q served to collect demographfic data, and to evaluate the severity of the disorder. On the day of the last stimulation, and one month after the last stimulation, subjects filled out the FCQ-S and the FCQ-T again.

Statistical package R, version 3.4.2 was used for the statistical processing of the data. The two-sample t-test method was used to compare the differences in cravings between subjects stimulated by the real and sham coils in all situations: before stimulation, directly after the last stimulation, and one month after the last stimulation. The paired t-test method was used to evaluate the changes of craving over time, meaning the difference in craving before the stimulation and on the last day of stimulation, and difference in craving on the last day of stimulation and one month after the last stimulation.

Parameters of stimulation A MAGSTIM Super Rapid 2 device with eight flat shaped coil was used to provide the rTMS. The control group was stimulated by a sham coil with similar side effects regarding sound and a pain perception on the scalp. The left DLPFC was chosen as the stimulation target. The coil placement for the DLPFC stimulation was 5 cm anterior in the same parasagital line from the place of maximum musculus abductor pollicis brevis response. The stimulation site was outlined on a cap, which was repositioned during each rTMS session.

The number of sessions was set on 10. Each stimulation session consisted of 15 trains of 10 s and 107 s intertrain, at a frequency of 10 Hz. That meant 1500 pulses applied during one session taking cca 20 minutes. The intensity of stimulation was 100% of minimal motor threshold (MMT). MMT was identified as the minimum magnetic field strength required to produce a motoric response of right thenar muscle, which was determined by visual control and controlled by EMG measurement. Stimulations were realized throughout a two week period, excepting weekends.

ELIGIBILITY:
Inclusion Criteria:

* having binge eating disorder
* being over the age of 18

Exclusion Criteria:

* contraindications for rTMS such as: a history of epileptic seizur paroxysms, increased intracranial pressure, brain tumor, implanted metal devices in the cranium (except the oral cavity), and any implanted peacemaker or drug pump
* non-compliance - inability to complet 10 sessions of stimulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The degree of craving | one month
  For evaluation of craving the Food Craving Questionnaire-State (FCQ-S) was used. The degree of craving was rated from "never" (0 points), through "rarely", "sometimes", "often", "usually", to "always" (5 points). The FCQ-State (FCQ-S) consisted of 15 questions, which are focused on the craving being dependent on the actual psychological conditions of the subject. The degree of craving can range from 0 to 65 points.
The degree of craving | one month
  For evaluation of craving the Food Craving Questionnaire-Trait (FCQ-t) was used. The degree of craving was rated from "never" (0 points), through "rarely", "sometimes", "often", "usually", to "always" (5 points). The FCQ-Trait (FCQ-T) consisted of 39 questions focused on the craving as a stable property over time. The degree of craving can range from 0 to 195 points.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baczynski TP, de Aquino Chaim CH, Nazar BP, Carta MG, Arias-Carrion O, Silva AC, Machado S, Nardi AE. High-frequency rTMS to treat refractory binge eating disorder and comorbid depression: a case report. CNS Neurol Disord Drug Targets. 2014;13(5):771-5. doi: 10.2174/1871527313666140307154823. PMID 24606720
- [Background] Nijs IM, Franken IH, Muris P. The modified Trait and State Food-Cravings Questionnaires: development and validation of a general index of food craving. Appetite. 2007 Jul;49(1):38-46. doi: 10.1016/j.appet.2006.11.001. Epub 2006 Dec 21. PMID 17187897
- [Background] Cepeda-Benito A, Gleaves DH, Fernandez MC, Vila J, Williams TL, Reynoso J. The development and validation of Spanish versions of the State and Trait Food Cravings Questionnaires. Behav Res Ther. 2000 Nov;38(11):1125-38. doi: 10.1016/s0005-7967(99)00141-2. PMID 11060941
- [Background] Downar J, Sankar A, Giacobbe P, Woodside B, Colton P. Unanticipated Rapid Remission of Refractory Bulimia Nervosa, during High-Dose Repetitive Transcranial Magnetic Stimulation of the Dorsomedial Prefrontal Cortex: A Case Report. Front Psychiatry. 2012 Apr 20;3:30. doi: 10.3389/fpsyt.2012.00030. eCollection 2012. PMID 22529822
- [Background] Gay A, Jaussent I, Sigaud T, Billard S, Attal J, Seneque M, Galusca B, Van Den Eynde F, Massoubre C, Courtet P, Guillaume S. A Lack of Clinical Effect of High-frequency rTMS to Dorsolateral Prefrontal Cortex on Bulimic Symptoms: A Randomised, Double-blind Trial. Eur Eat Disord Rev. 2016 Nov;24(6):474-481. doi: 10.1002/erv.2475. Epub 2016 Sep 15. PMID 27633286
- [Background] McClelland J, Bozhilova N, Nestler S, Campbell IC, Jacob S, Johnson-Sabine E, Schmidt U. Improvements in symptoms following neuronavigated repetitive transcranial magnetic stimulation (rTMS) in severe and enduring anorexia nervosa: findings from two case studies. Eur Eat Disord Rev. 2013 Nov;21(6):500-6. doi: 10.1002/erv.2266. PMID 24155247
- [Background] McClelland J, Kekic M, Bozhilova N, Nestler S, Dew T, Van den Eynde F, David AS, Rubia K, Campbell IC, Schmidt U. A Randomised Controlled Trial of Neuronavigated Repetitive Transcranial Magnetic Stimulation (rTMS) in Anorexia Nervosa. PLoS One. 2016 Mar 23;11(3):e0148606. doi: 10.1371/journal.pone.0148606. eCollection 2016. PMID 27008620
- [Background] Uher R, Yoganathan D, Mogg A, Eranti SV, Treasure J, Campbell IC, McLoughlin DM, Schmidt U. Effect of left prefrontal repetitive transcranial magnetic stimulation on food craving. Biol Psychiatry. 2005 Nov 15;58(10):840-2. doi: 10.1016/j.biopsych.2005.05.043. Epub 2005 Aug 8. PMID 16084855
- [Background] Van den Eynde F, Claudino AM, Mogg A, Horrell L, Stahl D, Ribeiro W, Uher R, Campbell I, Schmidt U. Repetitive transcranial magnetic stimulation reduces cue-induced food craving in bulimic disorders. Biol Psychiatry. 2010 Apr 15;67(8):793-5. doi: 10.1016/j.biopsych.2009.11.023. Epub 2010 Jan 8. PMID 20060105
- [Result] Jassova K, Albrecht J, Papezova H, Anders M. Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment of Depression and Anxiety in a Patient with Anorexia Nervosa. Med Sci Monit. 2018 Jul 30;24:5279-5281. doi: 10.12659/MSM.908250. PMID 30057403